CLINICAL TRIAL: NCT06838013
Title: A Randomized Controlled Trial of Anodal Transcranial Direct Current Stimulation and Transcutaneous Electrical Nerve Stimulation for Improving Lower Limb Function in Stroke Patients
Brief Title: Effect of Combining Central and Peripheral Cutaneous Electrical Stimulation on Lower Limb Motor Function in People With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023_GRF_Ng
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: transcranial direct current stimulation; transcutaneous electric nerve stimulation; stroke; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Anodal tDCS+Bi-TENS (Experimental): All subjects will receive eighteen 60-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: Transcranial direct current stimulation (tDCS); Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS); Behavioral: Lower-limb task-oriented training
- Sham-tDCS+Bi-TENS (Sham Comparator): All subjects will receive eighteen 60-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: Sham transcranial direct current stimulation (Sham-tDCS); Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS); Behavioral: Lower-limb task-oriented training
- Anodal tDCS+placebo-TENS (Placebo Comparator): All subjects will receive eighteen 60-minute sessions of intervention, 3 sessions per week for 6 weeks.
- Control training (Placebo Comparator): All subjects will receive eighteen 60-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: Sham transcranial direct current stimulation (Sham-tDCS); Device: Placebo transcutaneous electrical nerve stimulation (Placebo-TENS); Behavioral: Lower-limb task-oriented training

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — tDCS will be delivered by a constant-current electrical stimulator (DC-stimulator; Eldith, Ilmenau, Germany). Rectangular electrodes covered with a saline-soaked sponge will be used for the anode and cathode. The anode will be placed over the leg area of the motor cortex, on the lesioned side, with the medial border of the electrode placed laterally to Cz on the international electroencephalogram 10-20 system. The cathode will be placed above the contralateral orbit. The stimulation intensity will be set at 2 mA for 30 minutes.
  Arms: Anodal tDCS+Bi-TENS
Device: Sham transcranial direct current stimulation (Sham-tDCS) — Sham tDCS will be delivered by a constant-current electrical stimulator (DC-stimulator; Eldith, Ilmenau, Germany). Rectangular electrodes covered with a saline-soaked sponge will be used for the anode and cathode. The anode will be placed over the leg area of the motor cortex, on the lesioned side, with the medial border of the electrode placed laterally to Cz on the international electroencephalogram 10-20 system. The cathode will be placed above the contralateral orbit. The stimulation intensity will The stimulator will only be applied for the first and last 30 seconds.
  Arms: Control training; Sham-tDCS+Bi-TENS
Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS) — TENS will be delivered to the common peroneal nerve of both intact and paretic leg for 30 minutes using a 120z Dual-Channel TENS Unit (ITO Physiotherapy & Rehabilittaion, Co, Ltd, Tokyo, Japan). The TENS stimulation will be at 100 Hz, with 0.2 ms square pulses at an intensity of twice the sensory threshold (defined as the minimum intensity at which subject reported feeling a tingling sensation and below the motor threshold as indicated by the absence of muscle twitching.
  Arms: Anodal tDCS+Bi-TENS; Sham-tDCS+Bi-TENS
Device: Placebo transcutaneous electrical nerve stimulation (Placebo-TENS) — Placebo-TENS will be applied to identical-looking TENS devices, with the electrical circuit disconnected inside the devices. Placebo-TENS will be delivered to the common peroneal nerve of both intact and paretic leg for 30 minutes that set at 100 Hz, with 0.2 ms square pulses.
  Arms: Control training
Behavioral: Lower-limb task-oriented training — The lower-limb task-oriented training comprises 5 exercises for 30 minutes, namely stepping up and down, heel lift a dorsiflexed position, partial squatting, gait re-education and transition training.
  Arms: Anodal tDCS+Bi-TENS; Control training; Sham-tDCS+Bi-TENS

SUMMARY:
This study aims to evaluate the effectiveness of transcranial direct current stimulation (tDCS) and transcutaneous electrical nerve stimulation (TENS) in augmenting the efficacy of the lower limb task-oriented training in people with stroke. It is hypothesize that lower limb motor function can be best improved by combining anodal tDCS with TENS, when compared with sham-tDCS with TENS, anodal tDCS with placebo-TENS, or control training at improving ankle muscle strength, motor control of lower limbs, walking performance, functional mobility and community integration in people with stroke.

DETAILED DESCRIPTION:
The application of transcutaneous electrical nerve stimulation (TENS) over a paretic lower limb could augment the effects of task-oriented exercise therapy on lower limb motor function in people with stroke, possibly through increased excitability of sensorimotor cortex.

In transcranial direct current stimulation (tDCS), a weak electrical current is applied through electrodes placed on the scalp to modulate cortical excitability and neural activity in targeted brain regions. Anodal tDCS, specifically, involves positioning the positively charged electrode over the targeted cortical area, which facilitates neuronal depolarization and increases cortical excitability in the underlying brain tissue. The enhanced neural excitability induced by anodal tDCS could promote neuroplasticity and optimize motor learning processes, potentially through the modulation of N-methyl-D-aspartic acid (NMDA) receptor -dependent mechanisms and alterations in GABAergic activity, leading to improved motor function and rehabilitation outcomes in various neurological conditions.

The next question concerns whether anodal tDCS could be combined with TENS and whether their synergetic effects could maximise the motor output of paretic limbs in people with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. are between 50 and 85 years of age;
2. have had a single stroke more than 6 months and less than 15 years;
3. have at least 5 degrees of active ankle dorsiflexion in the antigravity position;
4. are able to walk 10 m independently, with or without a walking aid;
5. are able to score 6 or higher out of 10 on the abbreviated mental test;
6. have no skin allergies (e.g. redness or itchiness after application of the electrical stimulation pads) to electrical stimulation or electrodes;
7. are able to follow instructions and give informed consent.

Exclusion Criteria:

1. have any additional medical, cardiovascular or orthopedic conditions that would hinder their treatment or assessment;
2. have a cardiac pacemaker;
3. have aphasia or cognitive difficulties that may interfere with their comprehension of instructions;
4. have had one or more epileptic seizures within the year prior to the date of inclusion in the study;
5. have an intracerebral metal clip;
6. have a major somatosensory deficit
7. have any contraindication to tDCS;
8. are currently involved in drug studies or other clinical trials.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Paretic ankle dorsiflexor strength | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The paretic ankle dorsiflexor strength (in kilograms) is measured with a Nicholas hand-held dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN) in supine lying position. The muscle strength will be measured twice. The average strength of the 2 trials will be recorded. A higher value indicated a better paretic ankle dorsiflexor strength.
Paretic ankle plantarflexor strength | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The paretic ankle plantarflexor strength (in kilograms) is measured with a Nicholas hand-held dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN) in supine lying position. The muscle strength will be measured twice. The average strength of the 2 trials will be recorded. A higher value indicated a better paretic ankle dorsiflexor strength.
Fugl-Meyer Assessment of Lower Extremity (FMA-LE) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  FMA-LE is used to evaluate the lower extremity motor control, including reflexes, voluntary control of isolated movement and coordination. The scale score ranging from 0 to 34, with 17 items and ordinal scoring from 0 to 2. A higher score indicates a better lower extremity motor control.

SECONDARY OUTCOMES:
10-Meter Walk Test (10MWT) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The subject will be asked to walk 10 meter in a comfortable speed. The completion time will be records by stopwatch. The test will be repeated for 2 times. The completion time will be averaged. The shorter the completion time, the better performance is.
Timed 'Up and Go' test (TUG) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The TUG is used to measure the functional mobility. Each subject will be required to rise from a chair with armrests, walk 3 m forward, turn around, return to the chair and sit down. The time taken to complete this task will be measured in seconds with a stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged.
Lower-extremity motor co-ordination test | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The lower-extremity motor coordination test is used to measure the coordination of both the paretic and intact legs. Two red flat targets will be secured on the floor 30 cm apart. In sitting position with the feet resting flat on the floor and the heels on one of the targets, the participant will be instructed to touch 2 targets alternately with the big toe, as quickly and as accurately as possible, for 20 seconds. The number of times each target is touched will be counted. The more touch times indicated a better performance.
Gait Parameters (via GAITRite) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  Gait parameters will be assessed using the GAITRite system (CIR system, Inc., Havertown, Pennsylvania), a pressure-sensitive mat that automatically captures spatiotemporal gait characteristics. Participants will walk at their self-selected comfortable pace along the instrumented walkway.
Berg Balance Scale (BBS) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  BBS is a 14-item objective measure that assesses static balance and fall risk in adult patients. Items include tasks such as sitting to standing, standing unsupported, transfers, reaching, turning 360 degrees, and single-leg stance. Each item is scored from 0-4 points (0=unable to perform, 4=independent), with a maximum total score of 56 points. Higher scores indicate better balance.
Limits of Stability (LOS) Test | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The Limits of Stability (LOS) test quantifies participants' ability to intentionally shift their center of gravity (COG) to their stability limits without losing balance using Bertec Balance Advantage System (Bertec Corporation, Columbus, OH, USA). Participants stand on a force plate and shift their weight to move a cursor on a screen toward 8 targets arranged in a circular pattern at their theoretical limits of stability (100% LOS). Key parameters measured reaction time (RT) , movement velocity (MVL), directional control (DCL), endpoint excursion (EPE), maximum excursion (MXE). Higher scores indicate better dynamic balance control, except for reaction time where lower scores are better.
Sensory Organization Test (SOT) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  SOT assesses the participant's ability to maintain postural stability by evaluating the integration of visual, vestibular, and somatosensory inputs using Bertec Balance Advantage System (Bertec Corporation, Columbus, OH, USA). The test systematically disrupts sensory information while measuring postural sway.
  Outcome measures include composite equilibrium score and sensory analysis ratios (somatosensory, visual, vestibular, and preference ratios). Higher scores indicate better postural stability and sensory integration.
Cantonese version of Community Integration Measures (CIM-C) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item rating from 1 to 5 with a total score from 10 to 50. A higher CIM-C score indicates a higher level of community integration.
Foot & Ankle Disability Index Score (FADI) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  FADI is a 26-item patient-reported outcome measure that assesses functional limitations related to foot and ankle conditions. The questionnaire consists of 22 items assessing activities of daily living and 4 items specific to pain. Each item is scored on a 5-point Likert scale from 0 (unable to do) to 4 (no difficulty at all). Total scores are converted to percentages, with 100% representing no dysfunction. The FADI includes activities such as walking on even/uneven ground, climbing stairs, squatting, and recreational activities.
EQ-5D Visual Analogue Scale (EQ-5D VAS) | Baseline (0 week), Mid-intervention (3 weeks), Post-intervention (6 weeks), 1-month follow-up (10 weeks)
  The EQ-5D VAS is a standardized vertical visual analog scale (thermometer-like scale) that measures self-rated health status. Participants rate their overall health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state). This scale is part of the EQ-5D instrument but specifically captures the respondent's overall self-rated health status on the day of assessment. The VAS provides a quantitative measure of health outcome that reflects the participant's own judgment.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No